CLINICAL TRIAL: NCT01429571
Title: The Role of Antibiotics After Surgical Treatment of Simple Hand Infections: A Prospective Study
Status: Completed | Type: Observational
Sponsor: BG Trauma Center Tuebingen (Other)
Responsible Party: Principal Investigator, Dr. Theodora Manoli, MD, BG Trauma Center Tuebingen
Other Study IDs: Antibiotics in hand infections
Record Dates: First submitted 2011-09-01; First posted 2011-09-07 (Estimated); Last update posted 2011-09-07 (Estimated); Status verified 2011-09

CONDITIONS: Hand Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Systemic and local antibiotics
  Interventions: Other: No intervention
- Local antibiotics
  Interventions: Other: No intervention
- No antibiotics
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention
  Other Names: Since our study was observational after the beginning of treatment with or without antibiotics no intervention was influenced by the study.

SUMMARY:
Three patient groups with simple hand infections are tested regarding the necessity of antibiotics after surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with simple hand infections

Exclusion Criteria:

* Infection of the bone, tendon or joint
* Major diseases like diabetes or immunodeficiency
* Systemic manifestations like fever or lymphangitis
* Bite infections

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with simple hand infections (no infection of the bone, tendon or joint)
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- BG Trauma Center, Tübingen, Germany